

C.I. EOM-28-21

# CEIm Fundació Sant Joan de Déu

# DICTAMEN DEL COMITÉ DE ÉTICA DE LA INVESTIGACIÓN CON MEDICAMENTOS

Dra. Neus Riba Garcia Secretaria Técnica del CEIm Fundació Sant Joan de Déu

## **HACE CONSTAR:**

Que el CEIm Fundació Sant Joan de Déu en su reunión del 18/07/2024, acta 14/2024, ha evaluado la propuesta del promotor sobre la Modificación Sustancial nº 2 referida al estudio:

**Título:** "Estudio de hipersensibilidad a Anti-Inflamatorios No Esteroideos (AINES) en población pediátrica"

Investigador Principal: Adrianna Machinena Spera

Código CEIm: EOM-28-21

Servicio: Alergia e immunología clínica

Centro: Hospital Sant Joan de Déu - Esplugues HSJD.1 (FSJD)

## **Documentos con versiones:**

- Protocol. Versión 3, junio 2024.
- Hoja de información al paciente /padre o tutor legal. Versión 3, junio 2024.
- Hoja de consentimiento de los padres o tutor legal del menor participante
  (utilizar en estudios en los que participe un menor de 18 años). Versión 3, junio 2024.
- Hoja de información al paciente y asentimiento informado. Versión 3, junio 2024.

Que este CEIm considera que no se aumenta el riesgo de los pacientes y que se pueden cumplir las finalidades del estudio por lo que emite un **INFORME FAVORABLE** para la realización de la modificación anteriormente mencionada.

Que el CEIm Fundació Sant Joan de Déu, tanto en su composición, como en los PNT cumple con las normas de BPC (CPMP/ICH/135/95); se cumplieron los requisitos establecidos en la legislación vigente - Real Decreto 957/2020 - para que la decisión del citado CEIm sea válida; su composición actual es la siguiente:

### **Presidente:**

- Jesús Pineda Sánchez - Medicina – Pediatría

C.I. EOM-28-21 Página 1 de 2



C.I. EOM-28-21

# CEIm Fundació Sant Joan de Déu

### Vicepresidente:

Bernabé Robles Del Olmo - Medicina – Neurología

#### Secretaria:

- Neus Riba Garcia - Farmacología Clínica

#### **Vocales**:

- Fernando Aguiló Martínez Medicina Tropical
- Clara Chamorro Pérez Jurista
- Ángel del Campo Escota Representante de las asociaciones de pacientes
- Rosa María Dueñas Herrero Medicina Psiquiatría
- Pau Ferrer Salvans Farmacología Clínica
- María Eugènia Rey Abella Farmacia AP
- Ana Martín Ancel Medicina Neonatología
- Eduard Puig Vaquero Jurista Delegado protección de datos
- Carlota Romans Ruiz Farmacología Clínica
- Antoni Noguera Julián Medicina Pediatría
- Edurne Mazarico Gallego Medicina Ginecología y Obstetricia
- Esther Via Virgili Medicina Psiquiatría
- Oriol Martín Solé Medicina Cirugía y representante del CR
- Maite Gorostegui Obanos Medicina Oncología
- Rosa Farré Riba Farmacia hospitalaria
- Josep Codorniu Castelló Unidad Atención al Usuario
- Montserrat Gutierrez Juarez Enfermera

\*\*En el caso de que se evalúe algún proyecto del que un miembro sea investigador/colaborador, este se ausenta de la reunión durante la discusión del proyecto.

Para que conste donde proceda, y a petición del promotor,

Lo que firmo en Esplugues de Llobregat (Barcelona), a Fdo:

Dra. Neus Riba Garcia Secretaria Técnica del CEIm Fundació Sant Joan de Déu

C.I. EOM-28-21 Página 2 de 2